CLINICAL TRIAL: NCT02069821
Title: An Open-label, Multiple-dosing, Two-arms, One-sequence Study to Evaluate the Safety and Pharmacokinetics After Co-administration of Exforge® (Amlodipine Besylate/Valsartan) and Lipitor® (Atorvastatin Ca) in Healthy Male Volunteers
Brief Title: Pharmacokinetic Interactions Between Amlodipine Besylate/Valsartan and Atorvastatin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_EXA_101
Record Dates: First submitted 2014-02-19; First posted 2014-02-24 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): single administration : amlodipine/valsartan 10/160mg, qd, 10days(oral)
  Interventions: Drug: combination administration
- Group B (Experimental): single administration : atorvastatin 40mg, qd, 7days(oral)
  Interventions: Drug: combination administration

INTERVENTIONS:
Drug: combination administration — combination administration : amlodipine/valsartan 10/160mg and atorvastatin 40mg, qd, 10days(oral)

SUMMARY:
The purpose of the study is to assess the pharmacokinetic interactions between amlodipine besylate/valsartan and atorvastatin single or co-administered in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers in the age between 20 and 45 years old
2. The weight is over 55kg and is not exceed ±20% of ideal weight Ideal weight = [height -100]*0.9
3. Subjects with no history of any significant chronic disease
4. Judged to be in good health on the basis of routine laboratory data obtained prior to study drug administration
5. Willing to adhere to protocol requirements and sign a informed consent form

Exclusion Criteria:

1. Subjects with Symptoms of acute disease within 28days prior to study medication dosing
2. Subjects with a history of gastrointestinal diseases which might significantly change ADME of medicines
3. Subjects with a history of clinically significant allergies including drug allergies or anaphylaxis to amlodipine, valsartan and/or atorvastatin
4. Subjects with a history of myopathy
5. Subjects with a hereditary problems, for example, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
6. Subject with the mean blood pressure of siDBP ≥ 150 mmHg or ≤ 90 mmHg and/or siSBP ≥ 95 mmHg or ≤ 50 mmHg at the screening visit
7. Subjects with abnormal HDL-cholesterol(<35mg/dL)
8. Subjects with abnormal of serum potassium concentration (<3.4 mEq/L of >5.5 mEq/L in screening visit)
9. Subjects with a history of drug abuse
10. Subjects taking inducer or inhibitor of drug metabolism enzyme such as barbital within 28days prior to study medication dosing
11. Subjects who have received any drugs that might confound the results of the trial based on medical judgement by investigators within 14days prior to drug administration and OTC or vitamin within 7days prior to drug administration
12. Participated in a previous clinical trial within 60 days prior to dosing
13. Donated blood within 60 days prior to dosing
14. Subjects with a history of alcohol abuse(over 21 units/week, 1 unit = 10 g of pure alcohol) or is difficult to stop drinking within study
15. Subjects have ever smoked over 10 cigarette per day within 3 months prior to drug administration
16. Subjects with a history of caffeine abuse or or is difficult to stop drinking within study
17. Subjects with biliary obstruction
18. Subjects with hepatic dysfunction (AST or ALT >3 times to accepted normal range)
19. Subjects with moderate renal dysfunction (creatinine clearance (CLcr) < 30mL/min)
20. Subjects considered as unsuitable based on medical judgement by investigators

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To Evaluate PK interaction of amlodipine and valsartan | from pre dosing to 24hr post dose
  AUCss,τ, Css,max
To Evaluate PK interaction of atorvastatin and 2-OH atorvastatin | from pre dosing to 24hr post dose
  AUCss,τ, Css,max

SECONDARY OUTCOMES:
To Evaluate PK interaction of amlodipine and valsartan | from pre dosing to 24hr post dose
  tss,max, CLss/F, Css,min
To Evaluate PK interaction of atorvastatin and 2-OH atorvastatin | from pre dosing to 24hr post dose
  tss,max, CLss/F, Css,min

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam national university hospital, Daejeon, Jung-gu, South Korea

IPD SHARING:
Plan to Share IPD: No